CLINICAL TRIAL: NCT03413501
Title: A Multi-disciplinary Pain Intervention (MUD-PI) for Patients With Chronic Widespread Primary Pain
Acronym: MUD-PI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars-Petter Granan, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OsloUH Smerteklinikken
Record Dates: First submitted 2017-12-17; First posted 2018-01-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain, Widespread
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Receives treatment as usual at the clinic
- MUD-PI (Experimental): Receives multi-disciplinary pain intervention, agroup-based, multi-disciplinary treatment
  Interventions: Behavioral: MUD-PI

INTERVENTIONS:
Behavioral: MUD-PI
  Arms: MUD-PI

SUMMARY:
Patients who fulfilled inclusion criteria and consented to participate received either treatment as usual at the clinic, or were enrolled in a group-therapy based intervention, the multi-disciplinary pain intervention, led by a Medical doctor, physiotherapist and psychologist at the clinic.

DETAILED DESCRIPTION:
The Department of Pain Management and Research at Oslo University Hospital is Norway's largest outpatient pain clinic. It treats around one thousand new patients annually suffering from chronic pain of all aetiologies. Many of the patients receive interdisciplinary care based on a biopsychosocial framework, by at least two health care providers (physician, physiotherapist, psychologist, occupational therapist and/or nurse).

Participants were recruited through referrals from primary or secondary care, which were identified by an established interdisciplinary team. Patients found potentially eligible for the study were contacted by the research team and consulted with a research physician. Patients who fulfilled the inclusion criteria were invited to participate in the study and signed a consent form. Patients who declined to participate and non-eligible patients received usual care.

Inclusion criteria were 1) age 18 or more; 2) pain in at least three out of five bodily regions (defined as the four quadrants and axially); 3) pain persisting three months or more; 4) the patient was able to give informed consent and benefit from group therapy (including sufficient cognitive capacity and language skills); 5) no other medical condition could better explain the symptoms.

Subjects were randomised either to treatment as usual or a group-based multidisciplinary pain intervention (the MUD-PI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* Pain in at least three out of five bodily regions (defined as the four quadrants and axially)
* Pain persisting three months or more
* The patient was able to give informed consent and benefit from group therapy (including sufficient cognitive capacity and language skills
* No other medical condition could better explain the symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Change in Patient generated index | Change in score on inclusion and 1 week after completion of intervention or control group
  Individualised patient reported outcome

SECONDARY OUTCOMES:
Change in EQ-5D | Change in score on inclusion and 1 week after completion of intervention or control group
  standardised patient reported outcome
Change in Oswestry disability index | Change in score on inclusion and 1 week after completion of intervention or control group
  standardised patient reported outcome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschudi-Madsen H, Rodevand LN, Boymo Kaarbo M, Granan LP. Chronic Widespread Pain in a tertiary pain clinic: classification overlap and use of a patient generated quality of life instrument. Scand J Pain. 2019 Apr 24;19(2):245-255. doi: 10.1515/sjpain-2018-0097. PMID 30465720